CLINICAL TRIAL: NCT03651609
Title: Treatment for Ulnar Neuropathy at the Elbow - a Randomized Control Trial
Brief Title: Treatment for Ulnar Neuropathy at the Elbow
Acronym: UNETREAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Slovenian Research Agency (Other)
Responsible Party: Principal Investigator, Gregor Omejec, Principal Investigator, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNE Treatment
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Nervous System Diseases; Nerve Compression Syndromes; Cubital Tunnel Syndrome
Keywords: Ulnar neuropathy at the elbow; Electromyography; Ultrasonography; Treatment; Surgery; Conservative treatment
MeSH Terms: conditions — Peripheral Nervous System Diseases; Nerve Compression Syndromes; Cubital Tunnel Syndrome | interventions — Conservative Treatment

STUDY DESIGN:
Intervention Model Description: The study will have a parallel trial design with a 1:1 allocation ratio. CTE and RCC patients will be separately randomized throwing dice as follows: (1) even number - surgical release; and (2) odd number - conservative treatment. In patients with bilateral UNE, the more affected arm will be randomized. Patients randomized to the surgical arm will be referred to a plastic surgeon. All included CTE and RCC patients (including those randomized to surgical release) will be given illustrated instructions showing arm positions to avoid to prevent further ulnar nerve damage. The examiners will be blinded as far as possible to the patient's study arm and to the findings of other parts of the evaluation. Patients will not be blinded to treatment.
Who Masked: Investigator
Masking Description: Three examiners will perform one part of diagnostic evaluation that will include: (1) patients' history and focused neurological examination, (2) (EDx) and (3) US studies. They will be blinded to the findings of the other parts of the evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- UNE by CTE_surgery (Experimental): Patients with UNE by CTE randomly distributed for simple decompression of the ulnar nerve. Patients will also receive pictured recommendations with descriptions, which limb positions should be avoided. Control neurological examination will be performed every 3 months and identical protocol as at the time of diagnostic evaluation at 1 year follow-up.
  Interventions: Procedure: Simple decompression of the ulnar nerve; Behavioral: Conservative treatment
- UNE by CTE_conservative treatment (Active Comparator): Patients with UNE by CTE randomly distributed for conservative treatment. Patients will receive pictured recommendations with descriptions, which limb positions should be avoided. In order to prevent deterioration in conservatively treated group of patients with UNE by CTE control neurological examination will be performed every 3 months. Criteria for surgical release will be clinical deterioration or lack of clinical improvement after 12 months. Prior to surgical release and at 1 year follow-up identical protocol as at the time of diagnostic evaluation will be performed.
  Interventions: Behavioral: Conservative treatment
- UNE at RCC_surgery (Experimental): Patients with UNE at RCC randomly distributed for simple decompression of the ulnar nerve. Patients will also receive pictured recommendations with descriptions, which limb positions should be avoided. At 1 year follow-up identical protocol as at the time of diagnostic evaluation will be performed.
  Interventions: Procedure: Simple decompression of the ulnar nerve; Behavioral: Conservative treatment
- UNE at RCC_conservative treatment (Active Comparator): Patients with UNE at RCC randomly distributed for conservative treatment. Patients will receive pictured recommendations with descriptions, which limb positions should be avoided. At 1 year follow-up identical protocol as at the time of diagnostic evaluation will be performed.
  Interventions: Behavioral: Conservative treatment

INTERVENTIONS:
Procedure: Simple decompression of the ulnar nerve — Surgical release 2-3 cm distal to medial epicondyle with minimal-incision technique .
  Arms: UNE at RCC_surgery; UNE by CTE_surgery
Behavioral: Conservative treatment — Patients will be given pictured recommendations with descriptions, which limb positions should be avoided.

SUMMARY:
The purpose of the study is to investigate utility and appropriateness of treatment interventions taking into account the presumed mechanisms of two main varieties of ulnar neuropathy at the elbow (UNE). The investigators hypothesize that in patients with UNE by entrapment in the cubital tunnel (CTE) surgical release (simple decompression) is superior to conservative treatment. By contrast, in patients with UNE in the retrocondylar groove (RCC) surgical humero-ulnar apponeurosis (HUA) release (simple decompression) should not be superior to conservative treatment.

DETAILED DESCRIPTION:
Ulnar neuropathy at the elbow (UNE) is the second most common focal neuropathy with annual incidence rate of 21 per 100.000. Therefore, in Slovenia UNE each year affects approximately 420 and in Europe 156.000 patients. In previous publications evidence was presented that idiopathic UNE consists of two conditions occurring 2-5 cm apart. In the first condition, affecting about 15% of UNE patients, the ulnar nerve is entrapped 2-3 cm distal to the medial epicondyle (ME) in the cubital tunnel (CTE). In the second condition, affecting the majority (about 85%) of patients, the lesion is located at the ME or up to 4 cm proximally in the retrocondylar groove (RCC). As no anatomical structure constricting the ulnar nerve is usually found in that segment, the most probable cause of UNE at this location is extrinsic ulnar nerve compression against the underlying bone. The investigators believe that these two groups of UNE patients need different therapeutic approaches: (1) surgical release for ulnar nerve entrapment distal to ME and (2) conservative treatment for extrinsic nerve compression in the RCC. The efficiency of this therapeutic approach was already evaluated and significant clinical improvement was found in 80% of UNE patients. However, the design of that study did not enable to obtain an indisputable evidence that outcome was a result of treatment approach. It is still possible that improvement observed in patient population was a consequence of natural history rather than therapy. To resolve this problem a properly designed randomized control trial is needed. The investigators believe such trial would prevent numerous unnecessary and delayed operations in UNE patients.

ELIGIBILITY:
Inclusion Criteria:

* continuous numbness or paresthesias in the 5th ﬁnger,
* weakness of the ulnar-innervated muscles or hand clumsiness.

Exclusion Criteria:

* previous elbow fracture or surgery,
* polyneuropathy, symptoms of polyneuropathy, conditions causing polyneuropathy (e.g., diabetes) or multiple mononeuropathy,
* motor neuron disorders (e.g., monomelic amyotrophy, amyotrophic lateral sclerosis - ALS).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Podnar, MD, DSc, Principal Investigator — Department of Neurology, University Medical Center Ljubljana
Locations (1):
- University Medical Center Ljubljana, Department of Neurology, Institute of Clinical Neurophysiology, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification.
Supporting Information: Study Protocol, SAP
Time Frame: Already available, no end date.
Access Criteria: Anyone who wishes to access the data
URL: https://data.mendeley.com/datasets/s6mycc59v6/1

REFERENCES:
- [Background] Omejec G, Podnar S. Precise localization of ulnar neuropathy at the elbow. Clin Neurophysiol. 2015 Dec;126(12):2390-6. doi: 10.1016/j.clinph.2015.01.023. Epub 2015 Feb 14. PMID 25743266
- [Background] Omejec G, Podnar S. What causes ulnar neuropathy at the elbow? Clin Neurophysiol. 2016 Jan;127(1):919-924. doi: 10.1016/j.clinph.2015.05.027. Epub 2015 Jun 17. PMID 26093933
- [Background] Simon NG. Treatment of ulnar neuropathy at the elbow - An ongoing conundrum. Clin Neurophysiol. 2018 Aug;129(8):1716-1717. doi: 10.1016/j.clinph.2018.06.006. Epub 2018 Jun 18. No abstract available. PMID 29934265
- [Background] Omejec G, Podnar S. Long-term outcomes in patients with ulnar neuropathy at the elbow treated according to the presumed aetiology. Clin Neurophysiol. 2018 Aug;129(8):1763-1769. doi: 10.1016/j.clinph.2018.04.753. Epub 2018 Jun 1. PMID 29887400
- [Background] Omejec G, Zgur T, Podnar S. Diagnostic accuracy of ultrasonographic and nerve conduction studies in ulnar neuropathy at the elbow. Clin Neurophysiol. 2015 Sep;126(9):1797-804. doi: 10.1016/j.clinph.2014.12.001. Epub 2014 Dec 8. PMID 25541522
- [Background] Omejec G, Podnar S. Normative values for short-segment nerve conduction studies and ultrasonography of the ulnar nerve at the elbow. Muscle Nerve. 2015 Mar;51(3):370-7. doi: 10.1002/mus.24328. Epub 2015 Jan 10. PMID 24985195
- [Background] Omejec G, Podnar S. Proposal for electrodiagnostic evaluation of patients with suspected ulnar neuropathy at the elbow. Clin Neurophysiol. 2016 Apr;127(4):1961-7. doi: 10.1016/j.clinph.2016.01.011. Epub 2016 Jan 28. PMID 26971477
- [Background] Omejec G, Zgur T, Podnar S. Can neurologic examination predict pathophysiology of ulnar neuropathy at the elbow? Clin Neurophysiol. 2016 Oct;127(10):3259-64. doi: 10.1016/j.clinph.2016.08.002. Epub 2016 Aug 9. PMID 27552333
- [Background] Omejec G, Bozikov K, Podnar S. Validation of preoperative nerve conduction studies by intraoperative studies in patients with ulnar neuropathy at the elbow. Clin Neurophysiol. 2016 Dec;127(12):3499-3505. doi: 10.1016/j.clinph.2016.09.018. Epub 2016 Oct 13. PMID 27815973
- [Background] Omejec G, Podnar S. Neurologic examination and instrument-based measurements in the evaluation of ulnar neuropathy at the elbow. Muscle Nerve. 2018 Jun;57(6):951-957. doi: 10.1002/mus.26046. Epub 2018 Jan 23. PMID 29266317
- [Background] Podnar S, Omejec G, Bodor M. Nerve conduction velocity and cross-sectional area in ulnar neuropathy at the elbow. Muscle Nerve. 2017 Dec;56(6):E65-E72. doi: 10.1002/mus.25655. Epub 2017 Apr 15. PMID 28345147
- [Background] Leis AA, Smith BE, Kosiorek HE, Omejec G, Podnar S. Complete dislocation of the ulnar nerve at the elbow: a protective effect against neuropathy? Muscle Nerve. 2017 Aug;56(2):242-246. doi: 10.1002/mus.25483. Epub 2017 Jan 4. PMID 27859367

RESULTS

PARTICIPANT FLOW:
Groups:
- UNE at RGC_surgery: Patients with UNE at RGC randomly distributed for simple decompression of the ulnar nerve. Patients will also receive pictured recommendations with descriptions, which limb positions should be avoided. At 1 year follow-up identical protocol as at the time of diagnostic evaluation will be performed.
  Simple decompression of the ulnar nerve: Surgical release 2-3 cm distal to medial epicondyle with minimal-incision technique .
  Conservative treatment: Patients will be given pictured recommendations with descriptions, which limb positions should be avoided.
- UNE at RGC_conservative Treatment: Patients with UNE at RGC randomly distributed for conservative treatment. Patients will receive pictured recommendations with descriptions, which limb positions should be avoided. At 1 year follow-up identical protocol as at the time of diagnostic evaluation will be performed.
  Conservative treatment: Patients will be given pictured recommendations with descriptions, which limb positions should be avoided.
Period: Overall Study
Arm/Group | UNE by CTE_surgery | UNE by CTE_conservative Treatment | UNE at RGC_surgery | UNE at RGC_conservative Treatment
Started | 34 | 33 | 36 | 35
Completed | 32 | 33 | 33 | 32
Not Completed | 2 | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- UNE at RCC_surgery: Patients with UNE at RGC randomly distributed for simple decompression of the ulnar nerve. Patients will also receive pictured recommendations with descriptions, which limb positions should be avoided. At 1 year follow-up identical protocol as at the time of diagnostic evaluation will be performed.
  Simple decompression of the ulnar nerve: Surgical release 2-3 cm distal to medial epicondyle with minimal-incision technique .
  Conservative treatment: Patients will be given pictured recommendations with descriptions, which limb positions should be avoided.
- UNE at RCC_conservative Treatment: Patients with UNE at RGC randomly distributed for conservative treatment. Patients will receive pictured recommendations with descriptions, which limb positions should be avoided. At 1 year follow-up identical protocol as at the time of diagnostic evaluation will be performed.
  Conservative treatment: Patients will be given pictured recommendations with descriptions, which limb positions should be avoided.
- Total: Total of all reporting groups
Arm/Group | UNE by CTE_surgery | UNE by CTE_conservative Treatment | UNE at RCC_surgery | UNE at RCC_conservative Treatment | Total
Number analyzed (Participants) | 32 | 33 | 33 | 32 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 25 | 28 | 26 | 106
  >=65 years | 5 | 8 | 5 | 6 | 24
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [58 to 70] | 69 [59 to 72] | 58 [51 to 67] | 60 [51 to 66] | 63 [59 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 12 | 8 | 34
  Male | 25 | 26 | 21 | 24 | 96
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 32 | 33 | 33 | 32 | 130
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Slovenia | 32 | 33 | 33 | 32 | 130
Standard questionnaire for assessment of UNE severity (UNEQ) [Median (Inter-Quartile Range); unit: units on a scale] | 2.0 [1.8 to 2.3] | 2.0 [1.8 to 2.2] | 1.9 [1.8 to 2.0] | 1.9 [1.8 to 2.0] | 1.9 [1.8 to 2.1]

OUTCOME MEASURES:

1. Primary Outcome: UNEQ Score
Description: The primary outcome measure was the change in standard questionnaire for assessment of UNE severity (UNEQ) score from baseline at inclusion of patients into the study and at 12-month follow-up. The UNEQ considers the patient's numbness and tingling of the last two fingers, elbow pain, and changes in these symptoms with elbow position. It also evaluates hand weakness. Questionnaire items were graded as: 1 - absent, 2 - mild, 3 - moderate, 4 - severe, or 5 - very severe. The final UNEQ score was calculated as the mean of the nine items.
Time Frame: 1 year
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | UNE by CTE_surgery | UNE by CTE_conservative Treatment | UNE at RCC_surgery | UNE at RCC_conservative Treatment
Number analyzed (Participants) | 32 | 33 | 33 | 32
score on a scale
  Baseline | 2 [1.8 to 2.3] | 2 [1.8 to 2.2] | 1.9 [1.8 to 2] | 1.9 [1.8 to 2]
  12 monts | 1.7 [1.4 to 1.8] | 2 [1.8 to 2.1] | 1.4 [1.3 to 1.7] | 1.6 [1.3 to 1.7]

2. Secondary Outcome: Clinical UNE Severity
Description: Clinical UNE severity was graded: (1) Mild UNE - reduced sensation in the ulnar-innervated areas; (2) Moderate UNE - + ulnar hand muscle weakness, and (3) Severe UNE - + at least moderate ulnar hand muscle atrophy.
Time Frame: 1 years
Reporting Status: Not Posted, anticipated posting 2025-09

3. Secondary Outcome: Muscle Wasting
Description: The percentage of patients with reduction in ulnar-innervated hand muscle atrophy
Time Frame: 1 years
Reporting Status: Not Posted, anticipated posting 2025-09

4. Secondary Outcome: Muscles Strength
Description: The percentage of patients with increased ADM/FDI muscle MRC grade
Time Frame: 1 years
Reporting Status: Not Posted, anticipated posting 2025-09

5. Secondary Outcome: Light Touch 5th Finger
Description: Light touch sensation on the tip of the 5th finger as 0 - normal, 1 - moderately reduced, 2 - severely reduced or 3 - absent
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2025-09

6. Secondary Outcome: Ulnar_MNCV
Description: The percentage of patients with >30% increase in MNCVmin
Time Frame: 1 years
Reporting Status: Not Posted, anticipated posting 2025-09

7. Secondary Outcome: Ulnar_CMAP_AMP
Description: The amplitude of the ulnar CMAP on stimulation at D4
Time Frame: 1 years
Reporting Status: Not Posted, anticipated posting 2025-09

8. Secondary Outcome: Ulnar_SNAP_AMP
Description: The amplitude of the ulnar SNAP from the 5th finger
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2025-09

9. Secondary Outcome: Ulnar Nerve CSAmax
Description: ulnar nerve CSAmax in the elbow segment
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2025-09

10. Secondary Outcome: Ulnar Nerve CSAmin
Description: Ulnar nerve CSAmin in the elbow segment
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2025-09

ADVERSE EVENTS:
Time Frame: 2 years
Description: Patients reported adverse events at follow-ups. Additionally, principal investigator's phone number was given.
Arm/Group | UNE by CTE_surgery | UNE by CTE_conservative Treatment | UNE at RGC_surgery | UNE at RGC_conservative Treatment
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/33 | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/33 | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/33 | 0/33 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/09/NCT03651609/Prot_SAP_000.pdf